CLINICAL TRIAL: NCT05310006
Title: Acute Effects of Low and High-Speed Resistance Training on Blood Pressure in Older Adults: A Crossover Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Hélio José Coelho Júnior, Dr. Hélio José Coelho Júnior, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20021919
Record Dates: First submitted 2022-02-23; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Blood Pressure; Frailty
MeSH Terms: conditions — Frailty | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Speed Resistance Exercise (HSRE) (Experimental): Exercise sessions performed using eight times (sets) with 4-5 repetitions at 70-75% of the maximal strength. The concentric phase was performed as fast as possible, and the eccentric phase was carried out for 2 s.
  Interventions: Other: Exercise
- Traditional Resistance Exercise (TRE) (Experimental): Exercise sessions were performed using four sets of 8-10 repetitions at 70-75% of the maximal strength. The concentric and eccentric phases were carried out for 2 s.
  Interventions: Other: Exercise
- Control Session (CS) (No Intervention): Participants remained seated in a comfortable chair listening to music and/or talking with study investigators for approximately 30 min.

INTERVENTIONS:
Other: Exercise — Exercise sessions were performed in the morning (07:00 am-12:00 am) under the supervision of at least two fitness instructors in the rehabilitation unit of the nursing home.HSRE and TRE were designed according to the peculiarities of each type of resistance exercise (Chodzko-Zajko et al., 2009). During TRE, participants performed four sets of 8-10 repetitions at 70-75% of the maximal strength. The concentric and eccentric phases were carried out for 2 s. For HSRE, exercises were performed eight times (sets) with 4-5 repetitions at 70-75% of the maximal strength. The concentric phase was performed as fast as possible, and the eccentric phase was carried out for 2 s. Bilateral calf raise was performed using the same load as unilateral knee extension.
  Arms: High Speed Resistance Exercise (HSRE); Traditional Resistance Exercise (TRE)

SUMMARY:
The first study was a randomized crossover trial that compared the acute effects of High Speed Resistance Exercise (HSRE) and Traditional Resistance Exercise (TRE) on blood pressure parameters in a sample of frail older adults. Participants performed three experimental sessions (i.e., HSRE, TRE, and a control session [CS]) in a random order and separated from one another by seven days (standard deviation [±] 1 day). Food consumption was maintained constant during 48 h prior to the exercise session and a standard breakfast was offered 60-90 min before the beginning of the experimental sessions. The pharmacological therapy was kept constant during the whole study, and participants took their anti-hypertensive medication at the same time in all experimental days as prescribed by their physician.

ELIGIBILITY:
Inclusion Criteria:

- Aged ≥60 years; Frail according to Fried's criteria (Fried et al., 2009); Possessed sufficient physical and cognitive abilities to perform all exercises required by the protocol; Had a physician authorization to participate of exercise programs.

Exclusion Criteria:

Participation in a structured physical exercise training program in the past six months; Prescription of hormone replacement therapy and/or psychotropic drugs; Presence of any acute cardiovascular event (e.g., myocardial infarction) or complication in the past six months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Immediately after the end of the experimental sessions
  Blood Pressure
Blood Pressure | 10 minutes after the end of the experimental sessions
  Blood Pressure
Blood Pressure | 20 minutes after the end of the experimental sessions
  Blood Pressure
Blood Pressure | 30 minutes after the end of the experimental sessions
  Blood Pressure
Blood Pressure | 50 minutes after the end of the experimental sessions
  Blood Pressure
Blood Pressure | 60 minutes after the end of the experimental sessions
  Blood Pressure
Blood Pressure | 24 hours after the end of the experimental sessions
  Blood Pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Lar Mãe Mariana Nursing Home, Poá, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No